CLINICAL TRIAL: NCT03550963
Title: Research on Comparison Between Rice-richen Meal and Wheaten-richen Meal on Glucose Control Status Among Chinese Women With GDM
Brief Title: Comparison of Rice-richen and Wheaten-richen Meal on Glucose Control Among Chinese Women With Gestational Diabetes Melitus (GDM)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Liuyanping, Doctor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-1012
Record Dates: First submitted 2018-05-29; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy

STUDY DESIGN:
Intervention Model Description: All participants included in the study will be randomized assigned into one of two groups in parallel. Group one will be provided with rice-richen meal, while group two will be provided with wheaten-richen meal. All other factors, i.e. nutrition education, following-up, and physical activity will be the same between two groups.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rice-richen meal (Other): All participants included in the study will be randomized assigned into one of two groups in parallel, the rice-richen meal group and wheaten-richen meal group. The intervention of group one is that participants will be provided with rice-richen meal, meaning most of the calculated carbohydrates are from rice.
  Interventions: Other: rice-richen meal
- wheaten-richen meal (Other): All participants included in the study will be randomized assigned into one of two groups in parallel, the rice-richen meal group and wheaten-richen meal group.The intervention of group two is that participants will be provided with wheaten-richen meal, meaning most of the calculated carbohydrates are from wheaten.
  Interventions: Other: wheaten-richen meal

INTERVENTIONS:
Other: rice-richen meal — Participants in group one will be provided with rice-richen meal. All participants will be required to test and record blood glucose.
  Arms: rice-richen meal
Other: wheaten-richen meal — Participants in group two will be provided with wheaten-richen meal.All participants will be required to test and record blood glucose.
  Arms: wheaten-richen meal

SUMMARY:
Since the prevalence of gestational diabetes melitus (GDM) increased by ..., as an important part of medical treatment, nutrition therapy is highly required to help patients achieve normoglycemia. Carbohydrate intake is the primary nutrient affecting postprandial glucose levels,therefore the total amount and type of carbohydrate should be manipulated to blunt postprandial hyperglycemia. However,the type of carbohydrate has not yet been established. Rice and wheaten food have similar Glycemic Index (GI),but some researches found the glucose response to them is different. A case-control study is designed to compare the glucose control status between rice-richen meal and wheaten-richen meal, and all other macronutrients and micronutrients are all calculated and same between two groups, which may provide more clues for type of carbohydrate recommendation for Chinese women with GDM.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who undergo health examination in obstetric department in Peking Union Medical College Hospital.
* 20-45 years old.
* Pregnant women who are diagnosed with GDM according to the American College of Obstetricians and Gynecologists (ACOG) diagnostic criteria during 24-28 weeks.
* Be ability to use mobile medical equipment, conditional follow-up of the mother and child.
* Voluntary participation in this study.

Exclusion Criteria:

* Multiple pregnancy.
* Merger of serious diseases (such as hypertension, respiratory diseases, kidney disease, abnormal coagulation, immune system diseases, infectious diseases), history of adverse pregnancy (such as spontaneous abortion, habitual abortion), and history of GDM.
* Pregnant women with known diabetes before pregnancy, those requiring insulin or hormone therapy.
* Pregnant women who are deemed inappropriate to participate in this clinical study by her physician.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Study participants will be recruited from pregnant women who undergo health examination in Peking Union Medical College Hospital and meet the inclusion criteria.
Enrollment: 100 (Estimated)
Dates: Start 2018-06-23 (Estimated); Primary Completion 2018-11-23 (Estimated); Study Completion 2019-02-23 (Estimated)

PRIMARY OUTCOMES:
between-group difference in glucose control | 16 weeks
  comparison of the percentage of desired glucose status between two groups

SECONDARY OUTCOMES:
between-group difference in undesirable clinical outcome | 20 weeks
  comparison of incidence of macrosomia, dystocia, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Yanping Liu, master, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No